CLINICAL TRIAL: NCT05212987
Title: A Multi-center, Open, Single-arm Phase I Dose Exploratory Study to Evaluate the Safety, Tolerability, Pharmacokinetic Properties and Primary Antitumor Activity of FCN-098 in Patients With Advanced Solid Tumors
Brief Title: Study of FCN-098 in Patients With Advanced Solid Tumor
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fochon Pharmaceuticals, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FCN-098-001
Record Dates: First submitted 2021-12-28; First posted 2022-01-28 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2021-12

CONDITIONS: Solid Tumor
Keywords: Solid Tumor; NTRK

STUDY DESIGN:
Intervention Model Description: Open-Label Phase 1 Dose escalation study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose Escalation and Expansion (Experimental): FCN-098 will be given orally in ascending doses in patients with advanced solid tumor , until the maximum tolerated dose or recommended dose is reached.
  Interventions: Drug: FCN-098

INTERVENTIONS:
Drug: FCN-098 — FCN-098 will be given orally in ascending doses starting at 40 mg Q12h until the maximum tolerated dose or recommended dose is reached.

SUMMARY:
A multi-center, open, single-arm phase I dose exploratory study to evaluate the safety, tolerability, pharmacokinetic characteristics and primary antitumor activity of FCN-098 in patients with advanced solid tumors.

DETAILED DESCRIPTION:
This study is a multicenter, open, single-arm Phase I clinical study. The safety, tolerance and PK characteristics of FCN-098 in patients with advanced solid tumors were determined, the MTD of oral FCN-098 was determined, and the RP2D of FCN-098 was determined, and the efficacy of FCN-098 was preliminarily evaluated.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥ 18 years，no gender limitation；
* 2. Patients with inoperable solid tumors, stage III or IV, confirmed histologically or cytologically by standard treatment failure or no standard treatment;
* 3. Dose-escalation stage: patients with advanced solid malignancies after failure of standard treatment (patients with positive NTRK gene fusion or mutations in the TRK kinase region are preferred); Dose expansion stage: patients with advanced solid malignant tumors with NTRK gene fusion positive or TRK kinase region mutation after standard treatment failure; NTRK gene fusion positive or TRK kinase region mutation can be included based on the positive report of the local laboratory, but tissues must be provided to the central laboratory for confirmation;
* 4. The ECOG Scores 0 or 1 for physical fitness (Dose-escalation stage),0-2(Dose expansion stage);
* 5. Can understand and be willing to sign informed consent prior to the commencement of any research procedure;
* 6. Expected survival at least 12 weeks;
* 7. Patients with adequate organ and bone marrow function: absolute value of neutrophils ≥ 1.0 × 10^9/L (no G-CSF treatment within 7 days);Hemoglobin ≥ 80g/L (no erythrocyte infusion within 7 days);Platelet ≥ 75 × 10^9/L; Serum total bilirubin ≤ 1.5 × upper limit normal (ULN), and patients with Gilbert syndrome ≤3.0 × ULN. Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) ≤ 2.5 × ULN; For patients with liver metastasis, AST and ALT should be ≤ 5 × ULN. Creatinine<1.5×ULN or Creatinine clearance was ≥ 60 ml/min in dose-escalation stage, and ≥ 45ml/min in dose expansion stage. Creatinine clearance was calculated by Cockroft - Gault formula. Albumin ≥ 3g/dL;
* 8. At least one evaluable lesion (Dose escalation stage) was assessed according to RECIST 1.1 or RANO criteria; According to RECIST 1.1 or RANO standard to evaluate, at least one measurable lesions (Dose expansion stage) (primary central nervous system tumors according to the standard definition RANO, needs to have one or more measurable lesions by MRI assessment, size for at least 10 mm or more, and appeared in two or more ≤ 5 mm thick section, the measure does not include cystic cavity.) The imaging evaluation should be completed within 28 days before enrollment, and the patient's hormone dosage should be stable for at least 5 days or more.
* 9. A fertile woman must have a negative serum pregnancy test within 28 days of the first study drug administration and agree to contraception between 28 days before the first study drug administration and 90 days after the last study drug administration; Male patients are required to undergo ligation or agree to contraception and refuse sperm donation from 7 days before the first dose to 30 days after the last dose; The failure rate of contraceptive methods<1% per year, such as double screen contraceptive methods, condoms, oral or injectable contraceptives.

Exclusion Criteria:

* 1. Patients who received targeted therapy or tyrosine kinase inhibitor therapy within 2 weeks or within 5 half-lives (whichever is shorter) before starting administration, and who received chemotherapy, major surgery, radiotherapy, Anti-tumor biopharmaceutical treatment, immunotherapy or clinical trials within 4 weeks or within 5 half-lives (which is shorter);
* 2. Uncontrolled or symptomatic brain metastases (asymptomatic or stably controlled CNS metastases and no hormone therapy within 2 weeks are allowed to be enrolled);Patients with spinal cord metastasis with symptoms of spinal cord compression;Primary CNS tumors were allowed to be enrolled.
* 3. The toxicity of previous anti-tumor therapy has not recovered (>NCI-CITCAE 5.0 level 2), neurotoxic reaction level 2, except hair loss;
* 4. Patients should use strong CYP3A4 inhibitors (except drugs permitted in Section 6.8), inducers or sensitive substrates and sensitive substrates of CYP2B6, CYP2C8, CYP2C6 at the same time;
* 5. Patients take drugs (mainly Ia, Ic, class III anti-arrhythmia drugs) that will prolong the QTc interval or have risk factors for extending the QTc interval;
* 6. Difficulty in swallowing, or having an absorbance syndrome, or other medical conditions that prevent the absorption of drugs through the intestinal tract, or affect the absorption of FCN-098;
* 7. Cardiac function and disease meet one of the following conditions:

  1. screening period in research center 3 times of 12 lead ECG measurement, according to the instrument of QTc formula for calculating the average three times, QTc>470 ms for female and QTc>450 ms for male.
  2. continue uncontrolled hypertension, systolic blood pressure under antihypertensive treatment >150 mmHg, and/or diastolic pressure >100 mmHg.
  3. the American New York Heart Association (New York Heart Association, NYHA) classification of grade 3 or more congestive Heart failure;
  4. Arrhythmias of clinical significance, including but not limited to complete left bundle branch conduction anomaly, degree II atrioventricular block;
  5. within 6 months prior to screening of a history of heart attack or a stroke within three months.
* 8. Active bacterial, fungal or viral infections of clinical significance, including hepatitis B (hepatitis B virus surface antigen-positive with HBV DNA exceeding 1000 IU/ml or meet the criteria for active hepatitis B infection) or hepatitis C (HCV RNA positive), human immunodeficiency virus infection (HIV positive);
* 9. Suffered from a malignant tumor other than the selected indications in the past 5 years (other than fully treated cervical carcinoma in situ, non-melanoma basal cell or squamous epithelial cell skin cancer, local prostate cancer after radical operation, ductal carcinoma in situ after radical operation);
* 10. Women who are pregnant or breastfeeding. Any patient who becomes pregnant during the trial should withdraw from the study;
* 11.Rule out any situation that is not suitable for entry into the group. For example, it may cause confusion in research results, interfere with patients' participation in research procedures, or have a history of other diseases, treatments, or laboratory abnormalities, or current evidence that does not meet the clinical benefits of participating in the research. (Such as uncontrollable diabetes, active or uncontrollable infection, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2021-12-31 (Actual); Primary Completion 2024-05-08 (Estimated); Study Completion 2024-10-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicity within 2 days of single administration and 28 days of continuous administration. | From first dose up to 28 days
Determine the recommended phase II dose | From first dose up to 28 days

SECONDARY OUTCOMES:
To quantify the occurrence of adverse events (AEs) reported in all subjects who received study drug | From enrollment up to 30 days after last dose
  Incidence of untoward medical occurrences (adverse event = AE) in a participant who received study drug. Adverse events will be evaluated by dosing cohort and recorded according to NCI CTCAEv5 Common Toxicity Criteria.
To quantify the occurrence of TESAE during the treatment and cause permanent withdrawal of toxic effects | From enrollment up to 30 days after last dose
the death of the last medicine occurred within 30 days of frequency and cause of death | From enrollment up to 30 days after last dose
To quantify the Plasma Concentration of FCN-098 and its metabolite M1 (FCN-097) | 2 months
To determine the best overall response rate (ORR) by Response Criteria in Solid Tumors (RECIST) v1.1 in subjects with advanced solid tumors | Baseline up to approximately 1 year
  To evaluate the proportion of patients with an objective response (SD, PR, CR) as defined by RECIST 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Hu Xi chun, MD, Study Director — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No